CLINICAL TRIAL: NCT03560791
Title: A Review of Low-Dose CT Lung Cancer Screenings in a Community-Based Healthcare System With High Incidence
Acronym: REACH
Status: Completed | Type: Observational
Sponsor: St Elizabeth Healthcare (Other)
Responsible Party: Sponsor
Other Study IDs: 3/2018-022
Record Dates: First submitted 2018-05-07; First posted 2018-06-18 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An analysis of Low-Dose Cat Scan(LDCT) Screenings for Lung Cancer completed within the St. Elizabeth system from January 2015 until December 2019. The study investigator, or designee(s), will retrospectively review patient encounters, collecting data related to LDCT referrals and completions. Data analysis will focus on the subsequent imaging, procedures, reviews at The Nodule Review Board and Lung Cancers diagnosed as a result of the LDCT.

DETAILED DESCRIPTION:
This study is a single center, minimal risk, physician initiated retrospective chart review. Potential subjects will be identified using records provided by the St. Elizabeth Healthcare Thoracic Oncology and Radiology Department. Potential subjects will be screened for eligibility. Study investigator and designees will review patient electronic medical records, extracting data related to the ordering/completion of a LDCT and interventions that occurs thereafter. Collected data will focus on dates of encounters, diagnostic imaging/procedures, and treatments. Please see Appendix A for a complete list of data points. All of the data that will be collected for study purposes will be kept confidential. This will be attained by the following: First, each enrolled subject will be assigned a study specific serial number for the database. All study documents and data collection tools will be maintained with the investigative site file in a locked cabinet in a secure location maintained by the investigator. The database will not include the patient's name or hospital medical record number. No one will have access to the database but the study principal investigator and study staff designated by the principal investigator. However, study data may be reviewed by the Institutional Review Board of record, an appointed study monitor, an internal auditor for St. Elizabeth Healthcare, and necessary regulatory authorities. The security of the database will be maintained under the direction of the principal investigator. Fourth, when the study is completed, the manuscript is published, and IRB storage document requirements have been met, the file will be permanently deleted and destroyed

ELIGIBILITY:
Inclusion Criteria:

* Patients within St Elizabeth Healthcare who are referred for and/or have completed a LDCT from January 2015-February 2018
* >=18 years of age

Exclusion Criteria:

• Patient undergoes subsequent imaging, procedures and/or treatment at a facility outside of St. Elizabeth where records are not available through EPIC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients within St Elizabeth Healthcare who are referred for and/or have completed a LDCT from January 2015-February 2018
Sampling Method: Non-Probability Sample
Enrollment: 7659 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
Date(s) of LDCT | From patient referral for LDCT to completion of screening up to 1 year
  When the patient completed the LDCT(s)

SECONDARY OUTCOMES:
Additional Imaging caused by LDCTs | From patient referral through last radiographic image up to 6 years
Additional Procedures caused by LDCTs | From evidence of concerning nodule through completion of treatment up to 6 years
Adverse Events caused by LDCTs | From first screen through last treatment intervention for the nodule up to 6 years

OTHER OUTCOMES:
Nodule Categories | From first LDCT through final LDCT up to 6 years
Cancer Diagnosis | From detection of nodule through diagnostic pathology result up to 6 years
Stage of cancer diagnosis | From detection of nodule through diagnostic pathology result up to 6 years
Presentation in Tumor Board | From diagnosis of cancer through completion of treatment up to 6 years
Presentation in Nodule Review Board | From detection of category 4 nodule through completion of screening up to 6 years
Referral Date for LDCT | From identification of eligible patient through LDCT screen completion up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Royce Calhoun, MD, Principal Investigator — St Elizabeth Healthcare
Locations (1):
- St. Elizabeth Healthcare, Edgewood, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641